CLINICAL TRIAL: NCT00416169
Title: An Open Pilot Study to Evaluate the Safety and Efficacy of Galantamine in the Treatment of Pick's Disease/Frontotemporal Dementia /Pick Complex
Brief Title: A Pilot Study to Explore the Safety and Tolerability of Galantamine HBr in the Treatment of Pick Complex/Frontotemporal Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003106
Record Dates: First submitted 2006-12-22; First posted 2006-12-27 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Frontotemporal Dementia; Pick Complex
Keywords: Frontotemporal Dementia; Pick Complex; galantamine hydrobromide
MeSH Terms: conditions — Frontotemporal Dementia; Pick Complex | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine hydrobromide

SUMMARY:
The purpose of this study is to explore the safety and tolerability and the efficacy of galantamine treatment in subjects with Pick Complex/ Frontotemporal Dementia (PC/FTD). The safety and tolerability of galantamine therapy will be assessed over the entire treatment period (26 weeks). The 8 week withdrawal period will be used to confirm the safety of galantamine withdrawal in this subject group and it impact on any symptom improvement achieved during the first 18 weeks of galantamine treatment ( symptom improvement would be expected to stabilize or decline on withdrawal of an effective therapy).

The primary efficacy objective is to explore the effect of galantamine on behavior as measured by the Frontal Behavioral Inventory during the randomized withdrawal period. In addition, for subjects with primary progressive aphasia (limited ability for languages), the effects of galantamine on language will be explored using the Aphasia Quotient of the Western Aphasia Battery, and for all subjects the Clinical Global Impressions will be used to explore global change.

DETAILED DESCRIPTION:
Pick Complex (PC) and Frontotemporal Dementia (FTD) are a group of neurodegenerative dementias, initially characterized by frontotemporal lobar atrophy, that have overlapping clinical presentations and pathologic findings. Although the pathogenesis of Pick Complex/Frontotemporal Dementia remains unknown, and the neurotransmitter changes in Pick Complex/Frontotemporal Dementia are not well characterized, there is evidence for decreased cholinergic receptor binding in several cortical regions and decreased serotonin binding in the hypothalamus, frontal cortex, and temporal cortex. Galantamine is a reversible cholinesterase inhibitor. Recent studies indicate that galantamine is also an allosteric modulator at nicotinic cholinergic receptor sites. This nicotinic modulation appears to not only potentiate the response to acetylcholine binding, but also to modulate release of several other neurotransmitters, including serotonin. This pilot study will explore the safety and tolerability and efficacy of galantamine 8 mg and 12 mg twice a day treatment in subjects with Pick Complex/Frontotemporal Dementia. The study comprises an 18 week, open label, galantamine treatment phase followed by an 8 week, randomized, double blind, placebo controlled withdrawal phase. The safety and tolerability of galantamine therapy will be explored during both the open label and randomized withdrawal periods. The 8 week randomized withdrawal period will be used to confirm the safety of galantamine withdrawal in this subject group and its impact on possible symptom improvement achieved during the open label period as a marker for efficacy.

The expectation is that subjects who remain on galantamine for the additional 8 weeks will continue to improve or will remain stable with regard to their behavior, language, cognition, and global function, whereas subjects who are assigned to placebo will show a decline in some of these functions. This approach will allow an assessment of the effects of galantamine treatment (challenge) and galantamine withdrawal (de-challenge).

This study will involve a maximum of 40 subjects with Pick Complex/Frontotemporal Dementia. Subjects who meet the inclusion and exclusion criteria will receive galantamine 4 mg twice a day for 4 weeks followed by 8 mg twice a day for 4 weeks. At 8 weeks, the dose of galantamine will be maintained at 8 mg or increased to 12 mg twice a day based on tolerability. At the end of 12 weeks the dose of galantamine will be maintained at 8 or 12 mg twice a day or reduced to 8 mg twice a day, based on tolerability. The dose will be fixed for the remainder of the open label treatment period. Following 18 weeks of galantamine treatment, subjects will be randomly assigned (1:1) to continued treatment with galantamine (at the same dose) or placebo for an additional 8 weeks. Subjects and caregivers will be contacted by phone during the study and encouraged to contact the site at any time if they have concerns. If the subject's symptoms appear to be substantially worsening, and the investigator determines that the subject has deteriorated, he will advise the subject and caregiver about possible early completion of the study (early escape). Subjects electing early escape will complete final efficacy and safety assessments, then discontinue study medication. Once they have completed the study, they will begin the treatment of their choice in consultation with their physician. Subjects will be seen for assessment at Visit 1 (screening), Visit 2 (baseline), Visits 3 and 4 (12 and 18 weeks after the start of open label galantamine treatment), and Visit 5 (8 weeks after the start of the double blind withdrawal period or at early escape) or upon premature discontinuation. The subject and caregiver will return for an unscheduled visit if, in the judgment of the investigator, the subject requires clinical assessment between visits.

Subject selection criteria will ensure inclusion of subjects who have a clinical diagnosis of Pick Complex/Frontotemporal Dementia established by published consensus criteria and supported by neuroradiologic confirmation. The subjects selected for the study will have a diagnosis of primary progressive aphasia or frontotemporal dementia.

Safety and tolerability will be monitored by assessment of adverse events, electrocardiograms, physical examinations, blood pressure, heart rate, weight, and laboratory tests. Efficacy on symptoms will be explored by measuring changes in the Frontal Behavioral Inventory (FBI), the Aphasia Quotient (AQ) of the Western Aphasia Battery (WAB), the Mini Mental State Examination (MMSE), the Mattis Dementia Rating Scale (MDRS), the Frontal Assessment Battery (FAB), the Neuropsychiatric Inventory (NPI), the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Scale, the Clinical Global Impressions (CGI) Scales of Severity or Change, and subscales of the WAB and FBI. Changes in the results of neurologic examinations will also be documented.

The descriptive analyses will be performed, no hypotheses are specified for statistical testing. Safety and efficacy assessments will be summarized. Safety and Efficacy changes will be calculated from the screening/baseline of the galantamine treatment period to Week 18 (open label galantamine treatment period) and Week 26 (entire study for subjects randomized to galantamine for the 8 week withdrawal period). Comparisons between the placebo and galantamine treatment groups will use the changes in safety and efficacy parameters from Weeks 18 to 26 (the double blind, placebo controlled, randomized withdrawal period). Using a flexible dosing regimen, subjects will receive galantamine as oral tablets up to 8 or 12 mg twice per day for 18 weeks. Subjects will then be randomly assigned (1:1) in a double blind fashion to galantamine at the same dose or to placebo for an additional 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a clinical diagnosis of Frontotemporal Dementia or Pick Complex (PC/FTD) documented for at least 1 year with either primary progressive aphasia or frontotemporal dementia
* recent MRI or CT confirming frontotemporal lobar atrophy consistent with Frontotemporal Dementia or Pick Complex PC/FTD
* opportunity to perform certain activities of daily living as described in the Alzheimer's Disease Cooperative Study -- Activities of Daily Living Inventory
* living with or having regular visits (least 4 days/week) from a responsible caregiver
* Mini Mental State Examination score > 5 and the ability to complete baseline neuropsychometric testing
* able to see, hear, and communicate sufficiently, and willing to complete serial neuropsychometric tests
* female subjects of childbearing age must be surgically sterile or practicing an effective method of birth control before entry and throughout the study.

Exclusion Criteria:

* No neurodegenerative disorders and other causes of dementia or cognitive impairment from acute cerebral injuries, cerebrovascular disease or hypoxic cerebral damage, vitamin deficiency states, infection cerebral neoplasia
* no primary memory disturbance or an amnestic syndrome more compatible with Alzheimer's disease or other primary degenerative dementia
* no uncontrolled epilepsy or clinically significant psychiatric disease, cardiovascular disease, hepatic, renal, pulmonary, metabolic, or endocrine disturbances, active peptic ulcer and urinary outflow obstruction
* no use of any agent used for the treatment of dementia or other cognitive impairment
* no history of severe drug allergy or hypersensitivity to cholinesterase inhibitors, choline agonists or similar agents, or bromide

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-05; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
The safety is incidence of gastrointestinal events; efficacy are FBI, AQ and CGI. Changes will be calculated from baseline to Week 18 and Week 26. Comparisons between the placebo and galantamine groups will use the changes from Weeks 18 to 26.

SECONDARY OUTCOMES:
Secondary efficacy parameters are: MMSE, MDRS, FAB, NPI, ADCS-ADL Scale, subscales of the WAB and FBI and neurologic exams; safety are AE, ECGs, physical exam, vital signs, and lab tests.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A pilot study to evaluate the safety and tolerability of galantamine HBr in the treatment of Pick Complex/Frontotemporal Dementia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=503&filename=CR003106_CSR.pdf